CLINICAL TRIAL: NCT03875118
Title: Effects of Mouth-opening Training With Follow-up Telephone Calls on the Maximum Interincisal Opening and Mandibular Function of Postoperative Oral Cancer Patients: A Randomized Clinical Trial
Brief Title: Effects of Mouth-opening Training on the Maximum Interincisal Opening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Yuan's General Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20110818B
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Oral Cancer
Keywords: Oral cancer; Trismus; Mouth-opening training; Jaw exercise
MeSH Terms: conditions — Mouth Neoplasms; Trismus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Subjects in the intervention group received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks. Subjects in the intervention group received additional 6 follow-up phone calls (at 1, 2, 3, 4, 8 and 12-week after discharge) from the interventionist to enhance mouth-opening exercise adherence.
  Interventions: Behavioral: The mouth-opening training with follow-up telephone calls program
- The control group (Active Comparator): Subjects in the control group also received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks.
  Interventions: Behavioral: The mouth-opening training without follow-up telephone calls program

INTERVENTIONS:
Behavioral: The mouth-opening training with follow-up telephone calls program — Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks. Subjects in the intervention group received additional 6 follow-up phone calls (at 1, 2, 3, 4, 8 and 12-week after discharge) from the interventionist to enhance mouth-opening exercise adherence.
  Arms: The intervention group
Behavioral: The mouth-opening training without follow-up telephone calls program — Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks.
  Arms: The control group

SUMMARY:
PURPOSE:The purpose of the study was to investigate the effect of mouth-opening training with follow-up telephone calls for reducing postoperative trismus in patients with oral cancer.

METHODS:The study is a randomized clinical trial using repeated measures. Sixty-eight patients admitted at a general hospital in Taiwan for oral cancer surgery were recruited and randomly assigned to either the intervention or control group. All subjects were instructed to practice mouth-opening exercises three times a day every day for three months. Subjects in the intervention group received additional 6 follow-up phone calls to enhance mouth-opening exercise adherence. Data on maximum interincisal opening and mandibular function impairment were collected before surgery, at one-month, and three-months after discharge, using the TheraBite Range-of-Motion scale and Mandibular Function Impairment Questionnaire.

DETAILED DESCRIPTION:
The purpose of the study was to investigate the effect of mouth-opening exercise training with follow-up telephone calls for preventing postoperative trismus in patients with oral cancer. The specific aims were to test the intervention effects on enhancing mouth-opening exercise practice, MIO, and mandibular function. We hypothesized that the intervention group would show 1) better adherence to mouth-opening exercises, 2) greater MIO, and 3) better mandibular function over time, compared to the control group.

The study is a randomized clinical trial using repeated measures. A convenience sample of 68 oral cancer patients was recruited and randomly assigned to either the intervention or control group according to a list generated by the Random Allocation Software. Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks. Subjects in the intervention group received additional 6 follow-up phone calls (at 1, 2, 3, 4, 8 and 12-week after discharge) from the interventionist to enhance mouth-opening exercise adherence. Data on MIO and mandibular function impairment were collected before surgery, at one-month, and three-months after discharge, using the TheraBite Range-of-Motion scale and the Mandibular Function Impairment Questionnaire. The study was approved by the research ethics committee of the hospital where the data were collected.

All statistical analyses were carried out using the SPSS statistical package version 20.0 (SPSS Inc., Chicago, IL, USA). Characteristics of the subjects were summarized by percentages, means, and standard deviations (SDs). Chi-squared tests or Fisher's exact tests and two independent samples t-tests were used to examine group baseline equivalency. Value changes of study outcomes (MIO and mandibular function impairment) and mouth-opening exercises performed from T1, T2, to T3 were expressed in two study groups. A general linear model was used to model these outcomes as a function of main group effect and main time effect. An interaction term (group difference by time) was added into each model to investigate the synergistic effect of the intervention with time. Both the stability analysis and the analysis of repeated relationships were performed by generalized estimation equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older
2. diagnosed with oral cancer
3. scheduled for a primary curative oral cancer surgery
4. able to communicate in Mandarin or Taiwanese
5. obtained medical clearance from the patient's attending physician to participate in the study

Exclusion Criteria:

1. diagnosed with lip or tongue cancers which were less relevant to trismus
2. had central incisors extracted during the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Yuan's General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wetzels JW, Merkx MA, de Haan AF, Koole R, Speksnijder CM. Maximum mouth opening and trismus in 143 patients treated for oral cancer: a 1-year prospective study. Head Neck. 2014 Dec;36(12):1754-62. doi: 10.1002/hed.23534. Epub 2014 Jan 30. PMID 24478217
- [Background] Kamstra JI, van Leeuwen M, Roodenburg JLN, Dijkstra PU. Exercise therapy for trismus secondary to head and neck cancer: A systematic review. Head Neck. 2017 Nov;39(11):2352-2362. doi: 10.1002/hed.24859. Epub 2017 Jul 14. PMID 29044879
- [Background] Chen M, Li P, Lin F. Influence of structured telephone follow-up on patient compliance with rehabilitation after total knee arthroplasty. Patient Prefer Adherence. 2016 Mar 3;10:257-64. doi: 10.2147/PPA.S102156. eCollection 2016. PMID 27042020
- [Background] Agarwal P, Shiva Kumar HR, Rai KK. Trismus in oral cancer patients undergoing surgery and radiotherapy. J Oral Biol Craniofac Res. 2016 Nov;6(Suppl 1):S9-S13. doi: 10.1016/j.jobcr.2016.10.004. Epub 2016 Oct 22. PMID 27900243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to the hospital for curative oral cancer surgeries were recruited from surgical units of are going a teaching hospital in southernTaiwan. Potential subjects were referred by physicians and then screened by one of the researchers to determine their eligibility.
Pre-assignment Details: 72 people didn't meet inclusion criteria and 6 people decline to the study.
Groups:
- Mouth-opening Training With Follow-up Calls: Subjects in the intervention group received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks. Subjects in the intervention group received additional 6 follow-up phone calls (at 1, 2, 3, 4, 8 and 12-week after discharge) from the interventionist to enhance mouth-opening exercise adherence.
  The mouth-opening training with follow-up telephone calls program: Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks. Subjects in the intervention group received additional 6 follow-up phone calls (at 1, 2, 3, 4, 8 and 12-week after discharge) from the interventionist to enhance mouth-opening exercise adherence.
- Mouth-opening Training Without Follow-up Calls: Subjects in the control group also received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks.
  The mouth-opening training without follow-up telephone calls program: Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Subjects were instructed to practice the mouth-opening exercises three times a day, every day, for 12 weeks.
Period: Overall Study
Arm/Group | Mouth-opening Training With Follow-up Calls | Mouth-opening Training Without Follow-up Calls
Started | 34 | 34
Completed | 30 | 30
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mouth-opening Training With Follow-up Calls | Mouth-opening Training Without Follow-up Calls | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 47
  >=65 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  Taiwan | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: TheraBite Range-of-Motion Scale
Description: The TheraBite® Range-of-Motion Scale was used to measure the maximum incisal opening (MIO), which is the maximal vertical distance between the edges of the incisors of the maxilla and the mandible. The TheraBite® Range-of-Motion Scale is a disposable paper measuring scale specially designed to measure a subject's mouth and jaw opening. The subject sits in an upright position with his mouth open wide. For measuring the vertical opening, the scale has a possible range of 5 to 70 mm, with the notch is placed on the lower incisor midline. The usual range of MIO is between 40 and 55 mm. Subjects with MIO <35 mm are considered to have trismus.
Time Frame: Change from Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mouth-opening Training With Follow-up Calls | Mouth-opening Training Without Follow-up Calls
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 27.43 (10.71) | 26.57 (10.53)
  3 month later | 27.33 (9.73) | 16.17 (8.01)

2. Secondary Outcome: Mandibular Function Impairment Questionnaire (MFIQ)
Description: The MFIQ (Mandibular Function Impairment Questionnaire) was used to measure the extent of patients' mandibular function impairment. The questionnaire consists of 17 items, each of which targets a specific oral function impairment; including difficulties in social activity, speech, taking a large bite, chewing hard food, chewing soft food, work and/or daily activities, drinking, laughing, chewing resistant food, yawning, kissing, and eating different types of food. The subjects were asked to indicate how much difficulty they had with each activity or with eating each type of food using a 5-point Likert scale (0 = no difficulty, 4 = very difficult or impossible without help). The total score of the 17 items divided by 68 provides the scale score, with a possible range of 0 to 1. A higher score indicates greater severity of the mandibular function impairment. A score ≤ 0.3, between 0.3 and 0.6, and >0.6 indicates mild, moderate, and severe mandibular function impairment, respectively.
Time Frame: Change from Baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mouth-opening Training With Follow-up Calls | Mouth-opening Training Without Follow-up Calls
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 0.16 (0.21) | 0.17 (0.20)
  3 month later | 0.18 (0.23) | 0.55 (0.30)

ADVERSE EVENTS:
Time Frame: 3 month
Arm/Group | The Intervention Group | The Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Additional randomized controlled trials with longitudinal designs and larger sample sizes are needed to better define the role of the intervention in the treatment protocol for oral cancer associated trismus. Replicating this study in other settings is also recommended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes